CLINICAL TRIAL: NCT04929366
Title: Effects of Hemodialysis With Cooled Dialysate on High Sensitive Cardiac Troponin I (TnI) and Brain Natriuretic Peptide (NT proBNP)
Brief Title: Is Hemodialysis Associated With Cardiac Markers Change?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Osamah Hussein, Head of Internal Medicine A, Ziv Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0101-17-ZIV
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: End-Stage Kidney Disease; Hypothermic hemodialysis; Cardiovascular events; Troponin T; Brain natriuretic peptide
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-stage kidney patients treated in the dialysis unit group 1 (Experimental)
  Interventions: Procedure: Hypothermic dialysis followed with routine dialysis
- End-stage kidney patients treated in the dialysis unit group 2 (Experimental)
  Interventions: Procedure: Routine dialysis followed with hypothermic dialysis

INTERVENTIONS:
Procedure: Hypothermic dialysis followed with routine dialysis — Hypothermic dialysis (35.5 degrees Celsius dialysate) followed with routine dialysis (36.5 degrees Celsius dialysate)
  Arms: End-stage kidney patients treated in the dialysis unit group 1
Procedure: Routine dialysis followed with hypothermic dialysis — Routine dialysis (36.5 degrees Celsius dialysate) followed with hypothermic dialysis (35.5 degrees Celsius dialysate)
  Arms: End-stage kidney patients treated in the dialysis unit group 2

SUMMARY:
Hemodialysis (HD) triggers recurrent and cumulative ischemic insults to the brain and the heart. Cooled dialysate may have a protective effect on major organs and improve hemodynamic tolerability of dialysis. The aim of the study was to compare HD with cooled dialysate with routine dialysis in terms of hemodynamic stability and levels of high sensitivity Troponin I (hs-TnI) and N-terminal pro b-type natriuretic peptide (NTproBNP) post dialysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal insufficiency treated with dialysis for a period of at least three months.

Exclusion Criteria:

* Patients who experienced myocardial infarction during the three months prior to the start of the study
* Patients who underwent vascular surgery during the last month
* Patients who experienced chest pain at rest during the last week before the start of the trial - Patients who had to discontinue dialysis prematurely due to hemodynamic instability.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Comparison of hypothermic dialysis with routine dialysis in terms of hemodynamic stability | one year
  For each patient, four blood pressure measurements including systolic blood pressure, diastolic blood pressure and mean arterial pressure were performed at the beginning, after 2 hours, after 3 hours after 4 hours (end of hemodialysis).
Assessments of the levels of high sensitivite Troponin I (hs-TnI) and N-terminal pro b-type natriuretic peptide (NTproBNP) post dialysis | 6 months
  Blood samples were collected at the beginning of the dialysis session, and a second sample was taken in the last 5 minutes of hemodialysis in order to evaluate the relationship between hemodialysis with cooled dialysate (hypothermic dialysis) and the myocardial markers hs-TnI and NTproBNP and to monitor hypothermic hemodiaysis treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Younes Bathish, MD, Principal Investigator — Ziv Medical Centre, Safed, Israel / Azrieli Faculty of Medicine, Bar-Ilan University, Safed, Israel
Locations (1):
- Nephrology Department, Ziv Medical Center, Safed, Israel